CLINICAL TRIAL: NCT05525728
Title: Integrative Study of Vestibular Pathology With Analysis of Postural, Neurosensory, and Cognitive Disorders: Search for New Markers on the Causes and Consequences of Vertigo
Brief Title: Integrative Study of Vestibular Pathology
Acronym: SENSORIEL2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Stéphane BESNARD, Associate professor, University Hospital, Caen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-A02956-33
Record Dates: First submitted 2022-08-23; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Dizziness; Syndrome
Keywords: posture; vertigo; cognition; emotion; physiotherapist; vestibular system; balance
MeSH Terms: conditions — Dizziness; Syndrome; Vertigo

STUDY DESIGN:
Intervention Model Description: a group of patient suffering from vestibular pathology will be investigated regardless the etiology of the vertigo or dizziness
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient (Other): One cohort of patients
  Interventions: Other: Neurosensory

INTERVENTIONS:
Other: Neurosensory — Physiological and neurophysiological investigations

SUMMARY:
Exploratory posturological, neurosensory, cognitive, emotional, personality and general evaluations (quality of life).

The investigators will characterize a sensory profile quantified by one or more scores from a multi-parameter baysian approach. Each parameter and these scores will be correlated to the type of vestibular damage and its recovery in order to establish diagnostic, prognostic and therapeutic follow-up markers.

DETAILED DESCRIPTION:
This is an exploratory neurophysiological work that aims to identify diagnostic, prognostic and therapeutic markers in vestibular pathology.

Theinvestigators wish to characterize the neurosensory profile of individuals using new exploration paradigms provided by a new posturology platform coupled with virtual reality scenarios and by proposing a complete transversal approach in terms of evaluation of the subjects: personality, cognition, emotion including the depressive state, sensory strategy, general data.

Baysian statistical approaches and linear mixed model will be used to determine markers of sensory profile correlated to the vestibular damage for diagnostic, prognostic and therapeutic follow-up.

The investigators aim to be able to better characterize the cognitive-emotional and sensory deficits expressed by the vertiginous and unstable patients, to integrate it into the evaluation of the vestibular pathology, to use these markers to better discriminate the underlying physiopathological mechanisms, and to improve at the same time the diagnosis of the functional attack and the rehabilitation follow-up of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient (18-80 years old)
* Patient with an acute or chronic vestibular pathology according to ENT diagnostic criteria

Exclusion Criteria:

* Subjects under 18 years of age
* Pregnant or breastfeeding women,
* Persons in an emergency situation or unable to give their consent, including adults under guardianship
* Person under legal protection
* Patient presenting a vertigo or postural disorders of non vestibular etiology
* Persons deprived of liberty, minors, protected adults,
* Patients with an intercurrent neurological pathology including cerebellar pathology
* Inclusion of the subject in another interventional research protocol with pharmacological aim during the present study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-18 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Posture | through follow-up, an average of 6 months
  postural measurement
Cognition | through follow-up, an average of 6 months
  Spatial cognitive performance in a calibrated virtual radial maze
Personnality characteristic | through follow-up, an average of 6 months
  Evaluation of the BIg Five inventory test
Sleep | through follow-up, an average of 6 months
  Quantitative sleep recording
Emotion | through follow-up, an average of 6 months
  Anxiety measurement via questionnary

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Caen University Hospital, Caen
  - Frédéric Xavier, Vitrolles

IPD SHARING:
Plan to Share IPD: No